CLINICAL TRIAL: NCT05459987
Title: Feasibility and Impact of an Intensive Team-based Intervention on Prediabetes Remission in Patients With Coronary Heart Disease
Brief Title: Feasibility of Prediabetes Remission in Adults With Coronary Heart Disease
Acronym: DIABEPIC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Louis Bherer, Director of Centre EPIC research lab, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM 2022-3005
Record Dates: First submitted 2022-06-22; First posted 2022-07-15 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Prediabetic State; Coronary Heart Disease; Healthy Lifestyle; Remission
MeSH Terms: conditions — Prediabetic State; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Behavioral: Lifestyle changes Nutritional advice to progressively integrate a moderate-carbohydrate Mediterranean diet with intermittent fasting 16:8 (5 times/week for 12 weeks).
  Personalized exercise prescription and training (3 times per week)
  Personalized education and motivational interviewing
  Interventions: Behavioral: Lifestyle changes

INTERVENTIONS:
Behavioral: Lifestyle changes — Nutritional advice to progressively integrate a moderate-carbohydrate Mediterranean diet with intermittent fasting 16:8 (5 times/week for 12 weeks).
  Personalized exercise prescription and training (3 times per week)
  Personalized education and motivational interviewing

SUMMARY:
To evaluate the feasibility of a 6-month multidisciplinary program to reverse prediabetes in adults with coronary heart disease using the Mediterranean diet, intermittent fasting and exercise.

DETAILED DESCRIPTION:
The proposed study will assess the feasibility of an intensive lifestyle program to reverse newly onset prediabetes (HbA1c ≥ 5.7% to 6.4%) in patients with coronary heart disease that would otherwise start a standard cardiac rehabilitation programme (12 weeks with twice weekly exercise, nutrition, and nursing counselling). The patients will be offered an upgraded 6-month intensive team-based multidisciplinary stepwise program with the goal of remitting prediabetes. The program will consist of a 3-month synchronous nutritional, exercise, and motivational intervention and of a 3-month maintenance and follow-up period.

The DIABEPIC prevent 1 study is a single-arm, open-label study aiming to demonstrate the feasibility of an intensive multidisciplinary stepwise intervention in newly diagnosed prediabetic and coronary heart disease patients, ultimately aiming to remit prediabetes.

The purpose of this first study is to devise and iteratively improve participant recruitment and adherence strategies for a possible future randomized controlled trial. It also includes as goals: to study the efficacy and adherence of an intensive multicomponent lifestyle intervention, to study the proportion of patients that improve or remit their insulin resistant state, to study the changes in a variety of anthropomorphic, physical, analytic, vascular and test parameters and to better characterize the factors associated with prediabetes remission.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease patients referred from the Montreal Heart Institute.
* Aged ≥ 40 years.
* Recently diagnosed prediabetes (HbA1c ≥ 5.7% to 6.4%) in the last 6 months.
* Referred to Centre EPIC because of stable angina, acute coronary syndrome (with or without ST elevation), after coronary revascularization (primary or elective) or bypass surgery.
* Able to perform a maximal exercise test and exercise training program in accordance with current cardiovascular rehabilitation recommendations.
* Able to use a smartphone application or to complete an adherence/compliance diary.
* Able to read, understand and sign the information and consent form.

Exclusion Criteria:

* Absolute and relative contraindication to exercise testing and/or physical training.
* Diabetic patients (HbA1c ≥ 6.5%) or patients with a HbA1c value of ≥ 5.7% to 6.4% but with the help of oral hypoglycemic agents.
* Taking psychotropic medications that may induce mass gain (tricyclic antidepressants, mirtazapine, paroxetine, lithium, valproate, clozapine, olanzapine) or other medications known to promote mass gain (cortisone).
* Taking recently introduced weight-loss medications (semaglutide).
* Unintentional mass loss of more than 10 kg in the past year.
* Pregnant or nursing women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of an intensive multidisciplinary program based on lifestyle changes in coronary heart disease patients recently diagnosed with prediabetes that are referred to the Centre EPIC. | at 3 months after the start of the intervention
  Total recruitment, recruitment rate, compliance and completion rate at 3 months after the start of the intervention
Feasibility of an intensive multidisciplinary program based on lifestyle changes in coronary heart disease patients recently diagnosed with prediabetes that are referred to the Centre EPIC. | at 6 months after the start of the intervention
  Total recruitment, recruitment rate, compliance and completion rate at 6 months after the start of the intervention

SECONDARY OUTCOMES:
Proportion of prediabetic participants (HbA1c ≥ 5.7% to 6.4% at the start of the program) in complete remission of prediabetes. | at 3 and 6 months of the start of the intervention
  Remission of prediabetes will be defined by the following 3 criteria:
  1. An HbA1c < 5.7% at 3 months of intervention (Metabolic criteria).
  2. Which is maintained at 6 months (Duration criteria).
  3. Without the use of glucose-lowering agents (pharmacological criteria).
  Proportion of prediabetic patients that reach an HbA1c < 5.7% at 6 months of intervention will also be studied
Evolution of the HOMA-IR between the start of the program, the end of intervention (3 months) and the follow-up visit (6 months). | at 3 and 6 months of the start of the intervention
  HOMA-IR is a marker of insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
If sponsor OK, we would agree with making individual data available to other researchers
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: One year after completion of the study
Access Criteria: Upon request to the principal investigator

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Bommer C, Sagalova V, Heesemann E, Manne-Goehler J, Atun R, Barnighausen T, Davies J, Vollmer S. Global Economic Burden of Diabetes in Adults: Projections From 2015 to 2030. Diabetes Care. 2018 May;41(5):963-970. doi: 10.2337/dc17-1962. Epub 2018 Feb 23. PMID 29475843
- [Background] Hall KD, Ayuketah A, Brychta R, Cai H, Cassimatis T, Chen KY, Chung ST, Costa E, Courville A, Darcey V, Fletcher LA, Forde CG, Gharib AM, Guo J, Howard R, Joseph PV, McGehee S, Ouwerkerk R, Raisinger K, Rozga I, Stagliano M, Walter M, Walter PJ, Yang S, Zhou M. Ultra-Processed Diets Cause Excess Calorie Intake and Weight Gain: An Inpatient Randomized Controlled Trial of Ad Libitum Food Intake. Cell Metab. 2019 Jul 2;30(1):67-77.e3. doi: 10.1016/j.cmet.2019.05.008. Epub 2019 May 16. PMID 31105044
- [Background] Dal Canto E, Ceriello A, Ryden L, Ferrini M, Hansen TB, Schnell O, Standl E, Beulens JW. Diabetes as a cardiovascular risk factor: An overview of global trends of macro and micro vascular complications. Eur J Prev Cardiol. 2019 Dec;26(2_suppl):25-32. doi: 10.1177/2047487319878371. Epub 2019 Nov 13. PMID 31722562
- [Background] Lotta LA, Gulati P, Day FR, Payne F, Ongen H, van de Bunt M, Gaulton KJ, Eicher JD, Sharp SJ, Luan J, De Lucia Rolfe E, Stewart ID, Wheeler E, Willems SM, Adams C, Yaghootkar H; EPIC-InterAct Consortium; Cambridge FPLD1 Consortium; Forouhi NG, Khaw KT, Johnson AD, Semple RK, Frayling T, Perry JR, Dermitzakis E, McCarthy MI, Barroso I, Wareham NJ, Savage DB, Langenberg C, O'Rahilly S, Scott RA. Integrative genomic analysis implicates limited peripheral adipose storage capacity in the pathogenesis of human insulin resistance. Nat Genet. 2017 Jan;49(1):17-26. doi: 10.1038/ng.3714. Epub 2016 Nov 14. PMID 27841877
- [Derived] Iglesies-Grau J, Dionne V, Latour E, Gayda M, Besnier F, Gagnon D, Debray A, Gagnon C, Tessier AJ, Paradis A, Klai C, Martin N, Pelletier V, Simard F, Nigam A, L'Allier PL, Juneau M, Bouabdallaoui N, Bherer L. Cardiac Rehabilitation for Prediabetes and Metabolic Syndrome Remission: Impact of Ultraprocessed Food-Intake Reduction and Time-Restricted Eating in the DIABEPIC-1 Study. CJC Open. 2024 Aug 10;6(11):1411-1421. doi: 10.1016/j.cjco.2024.07.018. eCollection 2024 Nov. PMID 39582705
- [Derived] Iglesies-Grau J, Dionne V, Latour E, Gayda M, Besnier F, Gagnon D, Debray A, Gagnon C, Pelletier V, Nigam A, L'Allier PL, Juneau M, Bouabdallaoui N, Bherer L. Mediterranean diet and time-restricted eating as a cardiac rehabilitation approach for patients with coronary heart disease and pre-diabetes: the DIABEPIC-1 protocol of a feasibility trial. BMJ Open. 2023 Oct 17;13(10):e073763. doi: 10.1136/bmjopen-2023-073763. PMID 37848307